CLINICAL TRIAL: NCT07372794
Title: Electrical Impedance Tomography-Guided Respiratory Physiotherapy for Liberation From Prolonged Mechanical Ventilation: A Multicenter Randomized Controlled Trial
Brief Title: EIT-Guided Respiratory Physiotherapy for Prolonged Mechanical Ventilation (PMV)
Acronym: PMV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Yi Li, Principal Investigator, Senior Physiotherapist, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026bkky0115ly
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Prolonged Mechanical Ventilation; Respiratory Failure; Critical Illness
Keywords: Electrical Impedance Tomography; Prolonged Mechanical Ventilation; Respiratory Physiotherapy; Ventilator Weaning; Ventilator-Free Days
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-Guided Respiratory Physiotherapy (Experimental): Respiratory physiotherapy consists of airway clearance, chest physiotherapy techniques, breathing pattern optimization, and therapeutic positioning.
  In the EIT-guided group, real-time electrical impedance tomography (EIT) imaging is used during each physiotherapy session to individualize patient positioning and the selection and sequencing of physiotherapy techniques based on predefined ventilation distribution indicators.
  Interventions: Other: EIT-Guided Respiratory Physiotherapy
- Conventional Respiratory Physiotherapy (Active Comparator): Respiratory physiotherapy consists of airway clearance, chest physiotherapy techniques, breathing pattern optimization, and therapeutic positioning, delivered according to standardized institutional protocols without EIT guidance.
  Interventions: Other: Conventional Respiratory Physiotherapy

INTERVENTIONS:
Other: EIT-Guided Respiratory Physiotherapy — Respiratory physiotherapy consists of airway clearance, chest physiotherapy techniques, breathing pattern optimization, and therapeutic positioning, individualized using real-time EIT guidance based on predefined ventilation distribution indicators. Link this intervention to: Experimental Arm
  Arms: EIT-Guided Respiratory Physiotherapy
Other: Conventional Respiratory Physiotherapy — Respiratory physiotherapy consists of airway clearance, chest physiotherapy techniques, breathing pattern optimization, and therapeutic positioning, delivered according to standardized institutional protocols without EIT guidance. Link this intervention to: Control Arm
  Arms: Conventional Respiratory Physiotherapy

SUMMARY:
Patients with prolonged mechanical ventilation (PMV) frequently experience impaired ventilation distribution, respiratory muscle dysfunction, secretion retention, and delayed liberation from mechanical ventilation. Electrical impedance tomography (EIT) provides real-time bedside visualization of regional ventilation and enables individualized respiratory physiotherapy strategies.

This multicenter randomized controlled trial aims to evaluate whether EIT-guided respiratory physiotherapy improves ventilator-free days at day 28 compared with conventional respiratory physiotherapy in adult patients with PMV.

Respiratory physiotherapy consists of airway clearance, chest physiotherapy techniques, breathing pattern optimization, and therapeutic positioning. In the EIT-guided group, real-time EIT imaging is used to individualize physiotherapy strategies based on predefined ventilation distribution indicators, while the control group receives standardized physiotherapy according to institutional protocols without EIT guidance.

Secondary outcomes include successful liberation from mechanical ventilation, diaphragm ultrasound parameters, EIT-derived ventilation distribution indices (exploratory mechanistic outcomes), ICU Mobility Scale, healthcare resource utilization, and safety outcomes.

DETAILED DESCRIPTION:
This multicenter randomized controlled trial evaluates the effectiveness of electrical impedance tomography (EIT)-guided respiratory physiotherapy compared with conventional respiratory physiotherapy in adult patients with prolonged mechanical ventilation (PMV).

Eligible patients receiving invasive mechanical ventilation for at least 21 consecutive days will be randomly assigned in a 1:1 ratio to either the EIT-guided group or the control group, in addition to standard ICU care.

Respiratory physiotherapy consists of airway clearance, chest physiotherapy techniques, breathing pattern optimization, and therapeutic positioning. Both groups will receive standardized physiotherapy protocols with comparable treatment frequency and duration.

In the EIT-guided group, real-time EIT imaging will be used during each physiotherapy session. The control group will receive the same standardized physiotherapy components according to institutional protocols without EIT guidance.

The primary outcome is ventilator-free days at day 28 (VFD-28), defined as the number of days alive and free from invasive mechanical ventilation during the first 28 days after randomization. Patients who die before day 28 or remain invasively ventilated at day 28 will be assigned a value of zero. Reintubation within 72 hours will be considered treatment failure according to the predefined protocol.

Secondary outcomes include successful liberation from invasive mechanical ventilation by day 28, diaphragm ultrasound parameters, EIT-derived ventilation distribution indices (exploratory mechanistic outcomes), ICU Mobility Scale (IMS), healthcare resource utilization, and safety outcomes.

EIT-derived parameters are included as exploratory mechanistic outcomes to characterize physiological responses to the intervention and are not used for primary outcome adjudication.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Invasive mechanical ventilation for ≥ 21 consecutive days.
* Clinically stable and eligible for respiratory physiotherapy as determined by the treating team.
* Expected to remain on invasive mechanical ventilation for at least 48 hours after enrollment.
* Written informed consent obtained from the patient or legally authorized representative.

Exclusion Criteria:

* Contraindications to electrical impedance tomography .
* Hemodynamic instability requiring high-dose vasoactive support.
* Severe hypoxemia refractory to optimization.
* Unstable fractures or other contraindications to mobilization or positioning.
* Pregnancy.
* Expected death within 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days at Day 28 (VFD-28) | 28 days
  Ventilator-free days at day 28 (VFD-28) is defined as the number of days alive and free from invasive mechanical ventilation during the first 28 days after randomization. Patients who die before day 28 or remain invasively ventilated at day 28 will be assigned a value of zero. Reintubation within 72 hours after extubation or decannulation is considered treatment failure according to the predefined protocol.

SECONDARY OUTCOMES:
Successful liberation from invasive mechanical ventilation by day 28 | 28 days
  Successful liberation is defined as remaining free from invasive mechanical ventilation for at least 72 consecutive hours.
Diaphragm ultrasound parameters | Up to 28 days
  Diaphragmatic excursion, thickness, and thickening fraction measured by bedside ultrasound.
EIT-derived ventilation distribution indices | During intervention period (up to 28 days)
  Regional ventilation distribution indices derived from electrical impedance tomography, analyzed as exploratory mechanistic outcomes and not used for primary outcome adjudication.
ICU Mobility Scale (IMS) change from baseline | Up to ICU discharge or day 28
  Change in ICU Mobility Scale score from baseline to the highest achieved level during ICU stay.
ICU length of stay | Up to hospital discharge
  Number of days from ICU admission to ICU discharge.
Hospital length of stay | From hospital admission to hospital discharge
  Number of days from hospital admission to hospital discharge.
Total hospitalization cost | Up to hospital discharge
  Total direct medical cost during hospitalization.
Adverse events during physiotherapy | During intervention period (up to 28 days)
  Incidence of adverse events related to respiratory physiotherapy, including desaturation, hemodynamic instability, arrhythmia, or treatment intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Rehabilitation Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided